CLINICAL TRIAL: NCT07024459
Title: CARESCAPE Monitoring Systems ME Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11897644380
Record Dates: First submitted 2025-03-31; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-03

CONDITIONS: Surgery, Intensive Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- data collection (Experimental)
  Interventions: Device: Monitoring

INTERVENTIONS:
Device: Monitoring — Participants will be monitored with secondary monitor collecting data from parameters under evaluation

SUMMARY:
Improving the reliability and accuracy of the current parameter measurement technologies is always based on measurement data to develop a newer generation. Different parameters from different age groups will be studied under this study protocol.

DETAILED DESCRIPTION:
Improving the reliability and accuracy of the current parameter measurement technologies is always based on measurement data to develop a newer generation.

In this study it is essential to gain data from different age groups; children, adults, and elderly people since they are targeted population to use the devices in the future. In different age groups, there is e.g., a different physiological factures that may affect the product under development.

Different parameters will be studied under this study protocol. To get real picture of these parameters investigated, it is essential to also collect data from other parameters, e.g., electrocardiogram (ECG), oxygen saturation (SpO2) and carbon dioxide (CO2, including CO2 derived respiration rate (RR)).

The results of this study are intended to be used in product development purposes and as an additional data to support conformity to the general safety and performance requirements of the Medical Device Regulation within device's Clinical Evaluation process. The study described herein is being conducted to collect feedback from the parameters studied, and to collect the parameter raw data from the patients in the hospital units using the investigational devices.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent or have a Legally Designated Representative (LDR) to provide written informed consent;
2. Are being cared for in a hospital unit and are expected to remain in the unit for the duration of the study procedure; AND
3. Parameter(s) in scope of the study can be collected

Exclusion Criteria:

1. Are known to be pregnant;
2. Are breastfeeding;
3. Are suffering from infection(s) or immunocompromised patients that require isolation.
4. Have an implantable pacemaker if investigational parameters NMT and/or respiration rate are under evaluation
5. PI or designee decision due to subject's health condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of the performance and usability | From admission to discharge, maximum of 24 hours
  Primary outcome of this study is to conduct clinical evaluation of the performance and usability of the new software and hardware features introduced to the system by collecting data and surveys.

SECONDARY OUTCOMES:
Collection of data | From admission to discharge, maximum of 24 hours
  The secondary study outcome will be reached when the minimum number of subjects with good raw data quality have been collected and analyzed for product development.

OTHER OUTCOMES:
Collection of safety information | From admission to discharge, maximum of 24 hours
  Collection of number and type of AEs, SAEs and device issues

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Espoo, Uusimaa, Finland